CLINICAL TRIAL: NCT02200458
Title: Near-Infrared Software Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christie Medical Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP1019
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Vascular Access Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VeinViewer (Experimental): Vascular imaging technology will be used to visualize peripheral vasculature.
  Interventions: Device: VeinViewer

INTERVENTIONS:
Device: VeinViewer — Updated software on the VeinViewer device will be used to project an image of the vasculature on the skin.

SUMMARY:
This study will look at the performance capabilities of software for VeinViewer.

DETAILED DESCRIPTION:
This study will look at the performance capabilities of future software for VeinViewer.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age or older
2. Must be considered to be in overall good health by investigator
3. Must pass all prescreening questions
4. Must be able to read and understand English

Exclusion Criteria:

1. Presence of tattoos, scarring, and/or extensive hair in the areas to be assessed for cannulation.
2. IV cannulation in the arms or hands in the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Schears, MD, Principal Investigator — Christie Medical Holdings, Inc.
Locations (1):
- Christie Medical Holdings, Inc., Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VeinViewer: Vascular imaging technology will be used to visualize peripheral vasculature.
  VeinViewer
Period: Overall Study
Arm/Group | VeinViewer
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VeinViewer
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] — Average Age, Years
  Years | 37.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: CM] | 168.7 (10.5)
Weight [Mean (Standard Deviation); unit: kg] | 83.2 (17.6)
Fitzpatrick [Mean (Standard Deviation); unit: Points] — A numerical classification for human skin color: Type I (scores 0-6) Pale white, blond/red hair; blue eyes; freckles - Always burns/never tans. II (7-13) White/fair; blond/red hair; blue/green/hazel eyes - Usually burns/tans minimally. III (14-20) Cream white; fair with any hair/eye color; quite common - Sometimes mild burn/uniformly. IV (21-27) Olive to moderate brown; typical Mediterranean skin tone - Rarely burns/always tans well. V (28-34) Dark brown; South Asian skin types - Very rarely burns/tans very easily. VI (35+) Deeply pigmented dark brown to black - Never burns/tans very easily
  Points | 20.2 (7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Whom Successful Visualization of Vasculature Was Achieved
Time Frame: One day
Measure: Number; unit: participants
Arm/Group | VeinViewer
Number analyzed (Participants) | 62
participants | 62

ADVERSE EVENTS:
Arm/Group | VeinViewer
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes